CLINICAL TRIAL: NCT02442960
Title: An Open-Label, Dose-Escalation Phase Ib Study Evaluating the Safety and Preliminary Efficacy of Oral SA100 in the Treatment of Patients With Mild, Moderate or Severe Ulcerative Colitis
Brief Title: Evaluating Safety and Efficacy of Herbal Treatment in Ulcerative Colitis
Acronym: SA100
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30934
Record Dates: First submitted 2015-04-23; First posted 2015-05-13 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): Herbal treatment (SA100) 500 mg/day (250 mg twice per day)
  Interventions: Drug: Herbal treatment (SA100)
- Cohort 2 (Active Comparator): Herbal treatment (SA100) 1.5 g/day (750 mg twice per day)
  Interventions: Drug: Herbal treatment (SA100)

INTERVENTIONS:
Drug: Herbal treatment (SA100) — This treatment has been used extensively in traditional medicine practices for hundreds of years.
  Other Names: SA100

SUMMARY:
This is a 12-week, open-label, dose-escalation Phase 1b study of a herbal treatment given orally to subjects with ulcerative colitis. Subjects will be sequentially enrolled to one of two cohorts in up to two clinical sites. Treatment will be given for 8 weeks and study duration will be 12 weeks.

DETAILED DESCRIPTION:
This study consists of a 3-month period (12 weeks). You will receive study drug (SA100) for a 2-month period (8weeks) and then will continue to receive study assessements for an additional 1 month (4weeks). During the period in which you receive study drug (SA100), you will be asked to take the study drug twice a day (once in the morning and once in the evening), preferably at the same time each day. You will be assigned to one of three possible treatment groups. The three possible treatment groups are SA100 250 mg, 500 mg, or 750 mg. The group you are assigned to at the start of the study will remain the same throughout the study.

Blood samples, stool (feces), and tissue biopsies (up to 3 per region of colon) will be collected for testing purposes. These samples may also be kept for several years for future research.

An electrocardigram (ECG, which measures the electrical activity in your heart) will be taken at screening and week 2; and a flexible sigmoidoscopy will be performed at screening and week 8, (flexible tube that visualizes your intestine/colon and allows for tissue and stool to be obtained) to confirm your diagnosis of ulcerative colitis, to assess the severity of your disease, and for future testing of your tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 13 years and ≤ 75 years.
2. Mild, moderate and severe ulcerative colitis (biopsy-proven)
3. Mayo Scoring System Assessment of Ulcerative Colitis Activity score of 3 to 12 at screening.
4. Patients with active disease who are refractory to, intolerant to, or unwilling to take 5-aminosalicylic acid (5-ASA).
5. Patients of age ≥ 13 years and ≤ 17 years with active disease who are refractory or intolerant to 5-aminosalicyclic acid (5-ASA), corticosteroids, small molecule immunomodulators, and biologics or corticosteroid-dependent.
6. Physician's Global Assessment (PGA) Mayo subscore of at least 1 at screening.
7. Endoscopic evidence of active mucosal disease as assessed by flexible sigmoidoscopy with Mayo mucosal appearance subscore of at least 1 at screening.
8. Female patients of child-bearing potential must have a negative serum pregnancy test at the screening visit and agree to use two medically reliable methods of contraception (such as barrier with either spermicide or hormonal contraception) during the study period.
9. Male patients must be willing to use acceptable contraceptive methods and assure that their female partners of child-bearing potential use acceptable contraceptive methods during the study period.
10. Ability to adhere to the study visit schedule and other protocol requirements.
11. Adequate cardiac, renal, and hepatic function as determined by the principal investigators.
12. Written informed consent will be obtained before any study procedure is performed.

Exclusion Criteria:

1. Are nursing or pregnant.
2. Patients who are in critical condition
3. Crohn's disease or indeterminate colitis.
4. Known sensitivity to any ingredients in the study drug.
5. A change in therapy within 2 weeks before the baseline visit.
6. Use of immunomodulators (cyclosporine, mercaptopurine, azathioprine, etc.).
7. Diagnosis of diabetes, heart failure, unstable angina, liver or kidney disease, or any other unstable medical condition.
8. Any clinically meaningful laboratory abnormality that in the judgment of the investigator should preclude participation in the study.
9. Impaired renal function (serum creatinine levels >2.0 mg/dL) at screening.
10. Alanine transaminase (ALT) or aspartate transaminase (AST) laboratory values >1.5 times upper limit of normal at screening.
11. Diagnosis of Clostridium difficile, Salmonella, Shigella, Yersinia, Campylobacter, enteropathogenic E. coli in stool.
12. Positive test for hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg) at screening.
13. Active malignancy (except basal cell carcinoma).
14. Active alcohol or drug abuse.
15. Tobacco smoking within 2 weeks before study entry.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of herbal treatment (SA100) as assessed by clinical and laboratory adverse events. | Up to 12 Weeks
  To evaluate the safety and tolerability of oral SA100 given twice daily for 8 weeks, as assessed by clinical and laboratory adverse events.

SECONDARY OUTCOMES:
Total Mayo Score | Screening/Baseline, Week 8
  To evaluate preliminary efficacy (clinical response and remission rates) of oral SA100 based on (a) accepted disease activity and laboratory measures, including visual and histopathologic assessment of the colon by endoscopy, and (b) changes in serum biomarkers.
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | Screening/Baseline, Week 2, 4, 6, 8, 10, 12
  To evaluate preliminary efficacy (clinical response and remission rates) of oral SA100 based on (a) accepted disease activity and laboratory measures, including visual and histopathologic assessment of the colon by endoscopy, and (b) changes in serum biomarkers.
Biomarker levels (CRP & ESR) | Screening/Baseline, Week 8
  To evaluate preliminary efficacy (clinical response and remission rates) of oral SA100 based on (a) accepted disease activity and laboratory measures, including visual and histopathologic assessment of the colon by endoscopy, and (b) changes in serum biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Berkeley Limketkai, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Saiki JP, Andreasson JO, Grimes KV, Frumkin LR, Sanjines E, Davidson MG, Park KT, Limketkai B. Treatment-refractory ulcerative colitis responsive to indigo naturalis. BMJ Open Gastroenterol. 2021 Dec;8(1):e000813. doi: 10.1136/bmjgast-2021-000813. PMID 34969665